CLINICAL TRIAL: NCT00828854
Title: A Phase 2 Multicenter Study of the Effect of the Addition of SNDX-275 to Continued Aromatase Inhibitor (AI) Therapy in Postmenopausal Women With ER+ Breast Cancer Whose Disease is Progressing
Brief Title: Study of the Effect of the Addition of SNDX-275 (Entinostat) to Continued Aromatase Inhibitor (AI) Therapy in Postmenopausal Women With ER+ Breast Cancer Whose Disease is Progressing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0303
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: ER+ Breast Cancer
Keywords: breast cancer; estrogen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; Aromatase Inhibitors; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Entinostat 5 mg + AI (Experimental): Entinostat 5 mg tablet orally every week on Days 1, 8. 15 and 22 of each 28-day treatment cycle in combination with continued treatment with AI therapy at labeled dose and schedule until disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat; Drug: Aromatase Inhibitor (AI) Therapy

INTERVENTIONS:
Drug: Entinostat — Entinostat 5 mg PO every week
  Other Names: SNDX-275
Drug: Aromatase Inhibitor (AI) Therapy — AI therapy at labeled dose and schedule as prescribed in clinical practice. AI therapies include: Arimidex® (anastrozole) 1 mg/day by mouth (PO), Fermara® (letrozole) 2.5 mg/day PO , Aromasin® (exemestane) 25 mg/day PO.

SUMMARY:
The addition of entinostat to an AI will result in a maximal abrogation of estrogen receptor-α mediated activity and inhibit mechanisms of resistance to the aromatase inhibitor.

It is hypothesized that entinostat with continued AI will increase the estimated AI clinical benefit rate (CBR) from 5% to 25% with an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female patients.
2. Histologically or cytologically confirmed estrogen receptor-positive (ER+) breast cancer.
3. Progressive disease (PD) after at least 3 months on treatment with a 3rd generation AI in the advanced disease setting as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
4. At least 1 measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral computed tomography (CT) scan with the last imaging performed within 4 weeks prior to study entry. If there is only one measurable lesion and it is located in previously irradiated field, it must have demonstrated progression according to RECIST criteria.
5. Eastern Cooperative Oncology Group (ECOG) 0-1.
6. Laboratory parameters:

   1. Hemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x10^9/L; absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without the use of hematopoietic growth factors.
   2. Creatinine less than 2.5 times the upper limit of normal for the institution.
   3. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times the upper limit of normal for the institution.
7. Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

1. Discontinuation of AI therapy prior to study entry.
2. Less than 3 months treatment with most recent AI.
3. Rapidly progressive, life-threatening metastases, including any of the following:

   1. Symptomatic lymphangitic metastases.
   2. Patients with known active brain or leptomeningeal involvement.
4. More than one prior chemotherapy for metastatic disease.
5. Any chemotherapy within 3 months prior to study.
6. Radiotherapy to measurable lesion within 2 months prior to study.
7. Bisphosphonates initiated within 4 weeks prior to study start.
8. Allergy to benzamides or inactive components of study drug.
9. Previous treatment with entinostat or any other histone deacetylase (HDAC) inhibitor including valproic acid.
10. Patient is currently receiving treatment with any agent listed on the prohibited medication list such as valproic acid or other systemic cancer agents
11. Any concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases patient risk in the opinion of the investigator:

    1. Myocardial infarction or arterial thromboembolic events within 6 months, or experiencing severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease and a QTc interval >0.47 second.
    2. Uncontrolled heart failure or hypertension, uncontrolled diabetes mellitus, uncontrolled systemic infection,
    3. Other active malignancy within 5 years excluding basal cell carcinoma or cervical intraepithelial neoplasia [CIN / cervical carcinoma in situ] or melanoma in situ).
12. Patient currently is enrolled in (or completed within 30 days before study drug administration) another investigational drug study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2009-11-24 (Actual); Study Completion 2009-11-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- St. Vincent's University Hospital, Dublin, Ireland
- United Kingdom (5):
  - The University of Birmingham, Birmingham
  - Velindre Hospital - Whitchurch, Cardiff
  - Whiston Hospital; Clatterbridge Centre for Oncology, Liverpool
  - University College London Hospitals, London
  - Christie Hospital, Manchester Breast Centre, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United Kingdom and Ireland from 1 October 2008 to 24 November 2009.
Pre-assignment Details: Participants with a diagnosis of estrogen receptor-positive (ER+) breast cancer whose disease is progressing were enrolled to receive entinostat 5 mg in combination with continued aromatase Inhibitor (AI) therapy.
Period: Overall Study
Arm/Group | Entinostat 5 mg + AI
Started | 27
Completed (Completed=Completed Treatment) | 0
Not Completed | 27
Not completed — Disease Progression | 17
Not completed — Adverse Event | 9
Not completed — Reason not Specified | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set consisted of all eligible patients who signed informed consent.
Arm/Group | Entinostat 5 mg + AI
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  45 to 64 years | 7
  65 to 74 years | 15
  75 years and older | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 9
  United Kingdom | 18
Eastern Cooperative Oncology Group (ECOG) Status [Count of Participants; unit: Participants] — ECOG Performance status is an assessment of a participant's general well-being and activities of daily of life. Scores range from 0=perfect health (asymptomatic; able to carry out activities without restriction) to 5=death.
  Participants
    Score=0 | 9
    Score=1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants who achieved complete response (CR) or partial response (PR) or stable disease (SD) for 6 months as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started.
Time Frame: 6 months
Population: Per-protocol Set included participants from the full analysis who met eligibility criteria, completed at least 2 cycles and who had baseline and post-baseline tumor assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entinostat 5 mg + AI
Number analyzed (Participants) | 26
percentage of participants | 15.4 [4.4 to 34.9]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the number of months from the date of randomization to the earlier of progressive disease (PD) or death due to any cause.
Time Frame: Up to 6, 28-day cycles
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Entinostat 5 mg + AI
Number analyzed (Participants) | 26
months | 3.9 [1.9 to 5.6]

3. Secondary Outcome: Objective Response Rate (ORR) During the First 6 Cycles of Study Treatment
Description: ORR is defined as the percentage of participants with response during treatment classified as CR or PR, as assessed by the investigator based on RECIST, version 1.0. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 6, 28-day cycles
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entinostat 5 mg + AI
Number analyzed (Participants) | 26
percentage of participants | 3.9 [0.1 to 19.6]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Worsening of a pre-existing medical condition was considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. Abnormal clinical laboratory findings determined by the investigator to be clinically significant were recorded as AEs.
Time Frame: Up to 6, 28-day cycles + 30 days
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Entinostat 5 mg + AI
Number analyzed (Participants) | 27
Participants | 27

ADVERSE EVENTS:
Time Frame: Up to 6, 28-day cycles + 30 days
Description: Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | Entinostat 5 mg + AI
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entinostat 5 mg + AI (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Adverse drug reaction (General disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
VIth nerve paralysis (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entinostat 5 mg + AI (N=27)
Fatigue (General disorders) | 15
Nausea (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 13
Weight decreased (Investigations) | 11
Oedema peripheral (General disorders) | 10
Lethargy (Nervous system disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Pain (General disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Platelet count decreased (Investigations) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Chest pain (General disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Neutrophil count decreased (Investigations) | 4
Paraesthesia (Nervous system disorders) | 4
Urinary tract infection (Infections and infestations) | 4
White blood cell count decreased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 3
Depression (Psychiatric disorders) | 3
Dizziness (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood albumin decreased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Cellulitis (Infections and infestations) | 2
Depressed mood (Psychiatric disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eructation (Gastrointestinal disorders) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Lip dry (Gastrointestinal disorders) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Palpitations (Cardiac disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 2
Respiratory tract infection (Infections and infestations) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication